CLINICAL TRIAL: NCT00864370
Title: Bipolar Disorder in Pregnancy: Predictors of Morbidity
Brief Title: Bipolar Disorder (BPD) in Pregnancy: Predictors of Morbidity
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Massachusetts General Hospital (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Donald Jeffrey Newport, Associate Professor, Emory University
Other Study IDs: IRB00046058; R01MH071531 (NIH); Bipolar Disorder in Pregnancy (Other: Other)
Record Dates: First submitted 2009-02-25; First posted 2009-03-18 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Pregnancy; Bipolar Disorder
Keywords: Psychiatry; Pregnancy; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and urine samples are processed and stored at each research visit.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Very little is known about the impact of pregnancy and the postpartum period on BPD. As a result, the investigators have little evidence on which to base treatment guidelines. The main goal of this study is to help fill this gap by finding the risk factors for BPD relapse during pregnancy and the postpartum period.

The risk factors that the investigators will study include:

1. the severity of illness in the past
2. the type and severity of both recent and past stressors
3. any treatments received during pregnancy and the postpartum period.

Other goals of the study are:

1. to see what effect, if any, illness or any medicines taken during pregnancy have on the baby's well-being at delivery
2. to see how pregnancy alters the way the body clears any medicines taken for BPD
3. to see how much of these medicines babies are exposed to during pregnancy or breast-feeding.

The investigators believe that the information gathered in this study will lead to new treatment guidelines for BPD during pregnancy and the postpartum period that will improve outcomes for pregnant women with BPD and their babies.

DETAILED DESCRIPTION:
Despite the significant morbidity of bipolar disorder (BPD) and its high prevalence during the childbearing years, remarkably little is known about the impact of the female reproductive life cycle on BPD. Clinicians lack evidence-based guidelines for the perinatal management of BPD. The proposal addresses an understudied area with considerable public health implications for the estimated 100,000 women with BPD who conceive each year in the US.

The broad goal of this project is to delineate the clinical, psychosocial, and in particular, pharmacologic predictors of BPD recurrence during pregnancy. Preliminary findings suggest that inadequate treatment is a particularly robust predictor of prenatal BPD recurrence. Consequently, a specific emphasis will be placed on investigating the recurrence risk associated with suboptimal pharmacotherapy occurring as a result of medication discontinuation or declining drug concentrations secondary to increased prenatal clearance.

A prospective cohort design with monthly assessments will be implemented in a collaborative investigation between two of the leading perinatal psychiatry academic centers in the US with specific expertise in mood disorders research during pregnancy. The specific aims are 1) to quantify the risks for both syndromal and subsyndromal prenatal BPD illness associated with suboptimal pharmacotherapy while controlling for the severity of the previous course of illness and recent psychosocial stressors, 2) to examine the association of maternal prenatal BPD morbidity and psychotropic exposure with infant outcome at delivery thereby filling a current void and rounding out the requisite facets of the clinical risk/benefit assessment, and 3) to conduct pharmacokinetic (PK) modeling in an effort to delineate pregnancy-associated changes in drug clearance and provide initial reliable estimates of fetal drug exposure.

Study results will represent an incremental advance that: 1) elucidates risk factors for BPD morbidity during pregnancy; 2) contributes clinically relevant data to establish therapeutic guidelines for BPD during pregnancy; and 3) serve as a basis for preventive strategies aimed at optimizing maternal and infant outcome. Furthermore, the novel PK data will expand our understanding of prenatal drug metabolism, and the project will establish a cohort of children of women with BPD with detailed prospective prenatal histories.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy adult women (ages 18-45) fulfilling DSM-IV criteria for BPD of any subtype who are ≥ 16 weeks gestation dated by last menstrual period (LMP)
* Able to give informed consent and comply with study procedures

Exclusion Criteria:

* Actively suicidal or homicidal
* Active substance use disorder within 6 months prior to enrollment
* Positive urine drug screen
* Hematocrit < 30

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women of child bearing potential meeting DSM-IV (Diagnostic and Statistical Manual - IV) criteria for any subtype of Bipolar Disorder
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2005-05; Primary Completion 2011-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To determine if psychiatric morbidity among pregnant women with BPD is greatest for those who receive suboptimal pharmacotherapy, have a more severe past illness-course, or have experienced recent psychosocial stressors. | Nine months

CONTACTS AND LOCATIONS:
Overall Officials: D. Jeffrey Newport, MD, Principal Investigator — Emory Unviersity
Locations (1):
- Emory University Department of Psychiatry & Behavioral Sciences, Atlanta, Georgia, United States

REFERENCES:
- [Result] Newport DJ, Baldessarini RJ, Knight BT, Fernandez SV, Morris NJ, Viguera AC, Stowe ZN. Comparison of women with confirmed versus presumably misdiagnosed bipolar disorder. J Clin Psychiatry. 2012 Feb;73(2):242-6. doi: 10.4088/JCP.11m06936. Epub 2011 Dec 27. PMID 22225624
- [Result] Johnson KC, LaPrairie JL, Brennan PA, Stowe ZN, Newport DJ. Prenatal antipsychotic exposure and neuromotor performance during infancy. Arch Gen Psychiatry. 2012 Aug;69(8):787-94. doi: 10.1001/archgenpsychiatry.2012.160. PMID 22474072
- See also: Emory Women's Mental Health Program — http://womensmentalhealth.emory.edu/